CLINICAL TRIAL: NCT05466617
Title: Effects of a Gamified, Behavior Change Technique-Based Mobile App on Increasing Physical Activity and Reducing Anxiety in Adults With Autism Spectrum Disorder: Feasibility Randomized Controlled Trial
Brief Title: Gamified App on Increasing Physical Activity and Reducing Anxiety in Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American College of Sports Medicine Foundation (Unknown)
Responsible Party: Principal Investigator, Georgia Frey, Associate Professor Kinesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1807483245
Record Dates: First submitted 2022-07-11; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Autism Spectrum Disorder; Physical Activity; Anxiety; Mobile Health
MeSH Terms: conditions — Autism Spectrum Disorder; Motor Activity; Anxiety Disorders | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Two-group Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PuzzleWalk (Experimental): PuzzleWalk incorporates behavior change techniques (BCTs), a theory-based method of promoting healthy behavior change by leveraging psychological determinants. The example techniques included in PuzzleWalk are a comprehensive, visualized user guide, self-monitoring of target performance, contingent rewards, and goal setting.
  It is a spot the difference puzzle game comprising 660 major city images around the world. This format was chosen because it is easy to understand the purpose of the game, and it can quickly capture the user's interests without a complex comprehension process. Moreover, this visual image-based game facilitates visual interaction, which is a unique strength of individuals with ASD. The most unique design element of PuzzleWalk is the conversion algorithm between steps and game-solving time. Specifically, the user's accumulated steps are directly converted to game-solving time to motivate PA participation.
  Interventions: Behavioral: Mobile Health for Physical Activity Behavior Change
- Google Fit (Experimental): Google Fit (Google LLC) is a PA-tracking platform developed by Google for Android and Apple iOS. The app uses a sensor built into a smartphone device to automatically track PA, including steps and active minutes. It also allows users to journal and record a variety of forms of PA (eg, cycling, weightlifting, and yoga) by manually setting the activity tracking mode. Google Fit uses a heart point-based reward system as a gamification strategy to provide users with individualized exercise tips incorporated with PA recommendations outlined by the American Heart Association. The number of heart points received based on active minutes is the app's primary gamification strategy.
  Interventions: Behavioral: Mobile Health for Physical Activity Behavior Change

INTERVENTIONS:
Behavioral: Mobile Health for Physical Activity Behavior Change — All participants received visualized step-by-step instructions (eg, search and download on Google Play or App Store, user registration, goal setting, and PA behavior tracking) on the assigned PA app (PuzzleWalk or Google Fit) and used it from the beginning of the intervention start (fourth week) until the end of the intervention (eighth week). Both the PuzzleWalk and Google Fit groups received reminders regarding the use of the PA app during the first week of the intervention period and autonomously continued to use the app until the intervention ended.

SUMMARY:
Background: Physical activity (PA) has an impact on physical and mental health in neurotypical populations, and addressing these variables may improve the prevalent burden of anxiety in adults with autism spectrum disorder (ASD). Gamified mobile apps using behavior change techniques present a promising way of increasing PA and reducing sedentary time, thus reducing anxiety in adults with ASD.

Objective: This study aimed to compare the effectiveness of a gamified and behavior change technique-based mobile app, PuzzleWalk, versus a commercially available app, Google Fit, on increasing PA and reducing sedentary time as an adjunct anxiety treatment for this population.

Methods: A total of 24 adults with ASD were assigned to either the PuzzleWalk or Google Fit group for 5 weeks using a covariate-adaptive randomization design. PA and anxiety were assessed over 7 days at 3 different data collection periods (ie, baseline, intervention start, and intervention end) using triaxial accelerometers and the Beck Anxiety Inventory. Group differences in outcome variables were assessed using repeated-measures analysis of covariance, adjusting for age, sex, and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported medical diagnosis of anxiety or self-identification of experiencing anxiety symptoms for the past 3 or more months
* Access to a supported device (smartphones with Android 4.4 and higher or iOS 9.0 and higher operating system)
* Cognitive ability to understand the purpose of the study
* No prior experience using the PA mobile apps used in the study

Exclusion Criteria:

* Individuals with low cognitive function, co-occurring intellectual disabilities, or mobility impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Baseline Physical Activity and Changes from Baseline Physical Activity at 4th and 8th weeks | 7 days over three different data collection periods (total 21 days)
  Accelerometer-Measured Objective Physical Activity Levels

SECONDARY OUTCOMES:
Baseline Anxiety and Changes from Baseline Anxiety at 4th and 8th weeks | 7 days over three different data collection periods (total 21 days)
  Beck Anxiety Inventory (BAI; Beck, Epstein, Brown, & Steer, 1988) was used to assess participants' prolonged state of anxiety. The Beck Anxiety Inventory is a self-report scale comprising 21 items that measure the severity of anxiety symptoms during the past week. The score range is 0-63, with higher scores indicating greater degrees of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Frey, Ph.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee D, Frey GC, Cothran DJ, Harezlak J, Shih PC. Effects of a Gamified, Behavior Change Technique-Based Mobile App on Increasing Physical Activity and Reducing Anxiety in Adults With Autism Spectrum Disorder: Feasibility Randomized Controlled Trial. JMIR Form Res. 2022 Jul 28;6(7):e35701. doi: 10.2196/35701. PMID 35900808

DOCUMENTS (1):
  • Informed Consent Form (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT05466617/ICF_000.pdf